CLINICAL TRIAL: NCT05443009
Title: Evaluation of Self-Reported Pain in Children Submitted to Single Infiltration of Articaine During Primary Molar Extraction: Randomized Controlled Clinical Trial
Brief Title: Self-Reported Pain in Children Submitted to Single Infiltration of Articaine During Primary Molar Extraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Danielle Cristina Alves Rigo, Principal Investigator, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 030422
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Dental Pain; Anesthesia, Local
Keywords: articaine; lidocaine; child; pain
MeSH Terms: conditions — Toothache; Pain | interventions — Lidocaine; Carticaine

STUDY DESIGN:
Intervention Model Description: A blind, controlled, randomized, non-inferiority clinical trial with two parallel groups with allocation ratio will be 1:1
Who Masked: Outcomes Assessor
Masking Description: The evaluator will not know to which group the child belongs (anesthetic to be used), nor will he or she see the label of the anesthetic. He or she will be in the room during the initial anesthetic infiltration. All children will be considered participants in the control group, to conceal the anesthetic to be used. The evaluator will be asked to leave the room for as long as necessary to prevent learning whether or not the child receives an additional anesthetic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Active Comparator): Thirty-eight (38) children will receive conventional infiltration anesthesia (buccal infiltration injection followed by complementary injections on the palatal region) with 2% lidocaine and 1:100,000 epinephrine at a dose previously calculated by weight. Two-thirds of the anesthetic will be injected into the buccal area and 1/3 into the palatal area.
  Other Names: Control Group
  Interventions: Drug: Lidocaine
- Articaine (Experimental): Thirty-eightt (38) children will receive a single buccal infiltration injection with 4% articaine and 1:100,000 epinephrine at a dose previously calculated by weight.
  Other Names: Test Group
  Interventions: Drug: Articaine

INTERVENTIONS:
Drug: Lidocaine — A buccal infiltration injection followed by palatal injections and interpapillary injections of 2% lidocaine with 1:100,000 epinephrine will be administered.
  Other Names: Control Grup
  Arms: Lidocaine
Drug: Articaine — A single buccal infiltration injection of 4% articaine with 1:100,000 epinephrine will be administered.
  Other Names: Test Grup
  Arms: Articaine

SUMMARY:
The aim of this study is to analyze the effectiveness of articaine in controlling self-reported pain compared with conventional lidocaine anesthesia in children requiring extraction of deciduous maxillary molars. Only one extraction will be performed on each child. At least two consultations will be necessary to carry out the present controlled, randomized, and blinded study. All participants will be treated by the same dentist. Self-reported pain will be assessed using the Visual Analogue Scale.

DETAILED DESCRIPTION:
In the present study, self-reported pain during extraction of a maxillary primary molar with one buccal infiltration anesthesia with articaine will be compared with the conventional technique (buccal infiltration and palatal supplementation) with lidocaine. The study design will be a blind, controlled, randomized, non-inferiority clinical trial with two parallel groups. The anesthetic will be administered according to the weight of the child, using a table with the amount of anesthetic per weight group and the maximum recommended dose as reference. The hypothesis is that articaine, due to its anesthetic properties, is able to anesthetize as well as lidocaine with only one oral infiltration, without the need for additional anesthesia, which may guarantee better participant comfort, less dental anxiety, and less chair time. The use of the Visual Analogue Scale is important to assess the pain perceived by the children and to ensure the reliability of the responses. Participant comfort will be evaluated at each stage of the proposed treatment, and withdrawal from participation will be guaranteed at any time.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria: the presence of coronary destruction precluding restoration or adequate use of absolute isolation for endodontic and restorative procedures; perforation of the pulp chamber floor.
* Radiographic criteria: deciduous molars with at least one non-resorbed half-length root presenting carious lesions or defective restorations associated with signs or symptoms suggestive of pulp necrosis with endodontic contraindication (periapical or interradicular lesion extending over more than half of the roots or involving the crypt of the permanent successor tooth; the presence of pathologic resorption of more than 1/3 of one or more roots; failure of endodontic treatment with the persistence of periapical or inter-radicular lesion with or without clinical signs and symptoms; internal resorption).

Exclusion Criteria:

* Participants with acute pain or presence of odontogenic infection associated with systemic signs and symptoms and in cases of urgency;
* History of bleeding or blood clotting problems or taking medications that alter blood clotting prior to the procedure;
* Hypersensitivity or history of allergy to the drugs used in the research;
* Asthma;
* History of liver disease;
* History of sulfite allergy;
* Report of post-traumatic stress disorders or recurrent hospitalizations, personality or anxiety disorders, diagnosis of phobias or definite uncooperative behavior;
* Neurological disorders or communication difficulties;
* Use of analgesic or anti-inflammatory medications up to 5 hours before the procedure;
* Parents or guardians unable to be available for follow-up and/or respond to information necessary for the survey within 24 hours of the procedure.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Dental Pain | Immediately after the maxillary primary molar extraction
  Self-assessment of pain using the Visual Analogue Scale (VAS 0-100mm, higher values represent a worse outcome)

OTHER OUTCOMES:
Dental Pain | During the injection of local anesthesia and the surgical procedure
  Pain is evaluated by the outcome assessor using the Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale (FLACC 0-10 score, higher values represent a worse outcome) and the Faces Pain Scale - Revised (FBRS 0-10 score, higher values represent a worse outcome)
Dental Pain | Immediately after the injection of local anesthesia and the maxillary primary molar extraction
  Self-assessment of pain using the Wong-Baker FACES Pain Rating Scale (FACES 0-10 score, higher values represent a worse outcome)
Dental Pain | Immediately after the injection of local anesthesia
  Self-assessment of pain using the Visual Analogue Scale (VAS 0-100mm, higher values represent a worse outcome)
Heart rate variability | Immediately before, durin, and immediately after the surgical procedure
  Heart rate variability to be verified and recorded with the heart rate sensor (Polar H-10)
Heart rate | Immediately before, durin, and immediately after the surgical procedure
  Heart rate to be verified and recorded at moments described above carried out with the heart rate sensor (Polar H-10) and pulse oximeter
Evaluation of Post-surgical Pain | 24 hours after the surgical procedure
  Self-assessment of pain using a Visual Analogue Scale (VAS 0-100 mm, higher values represent a worse outcome) and the Faces Pain Scale - Revised (FBRS 0-10 score, higher values represent a worse outcome) in the postoperative period. It will be applied through teleconsultation

CONTACTS AND LOCATIONS:
Overall Officials: Mariane Cardoso, PhD, Study Director — Universidade Federal de Santa Catarina - UFSC; Carla Santana, PhD, Study Director — Universidade Federal de Santa Catarina - UFSC
Locations (4):
- Brazil (4):
  - Centro de Especialidades Odontológicas (CEO), Florianópolis
  - Centro de Especialidades Odontológicas (CEO), Palhoça
  - Universidade Federal de Santa Catarina - USFC, Santa Catarina
  - Centro de Especialidades Odontológicas (CEO), São José

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tirupathi SP, Rajasekhar S. Can single buccal infiltration with 4% articaine induce sufficient analgesia for the extraction of primary molars in children: a systematic literature review. J Dent Anesth Pain Med. 2020 Aug;20(4):179-186. doi: 10.17245/jdapm.2020.20.4.179. Epub 2020 Aug 27. PMID 32934983
- [Background] Taneja S, Singh A, Jain A. Anesthetic Effectiveness of Articaine and Lidocaine in Pediatric Patients During Dental Procedures: A Systematic Review and Meta-Analysis. Pediatr Dent. 2020 Jul 15;42(4):273-281. PMID 32847666
- [Derived] Rigo DCA, Santos PS, Moccelini BS, Rocha AO, Garcia JM, Ramos I, Santana CM, Cardoso M. Self-reported pain after buccal infiltration of articaine vs buccal and palatal infiltration of lidocaine for maxillary primary molar extractions: A noninferiority randomized clinical trial. J Am Dent Assoc. 2025 Nov;156(11):909-919. doi: 10.1016/j.adaj.2025.07.014. Epub 2025 Sep 11. PMID 40932429